CLINICAL TRIAL: NCT02555072
Title: Yellow Fever Vaccine Immunity After 1 Dose of Vaccine in Children and Adults: a Cohort Study in Non-endemic Area
Brief Title: Immunity Period After One Dose of Yellow Fever Vaccine in Adults and Children (Paraiba Study)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ASCLIN 005/2014
Record Dates: First submitted 2015-04-22; First posted 2015-09-21 (Estimated); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Yellow Fever Vaccine; Immunity
Keywords: Yellow Fever Vaccine, immunity evolution
MeSH Terms: interventions — Yellow Fever Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- naive children and adults for yellow fever vaccine (Other): both sexes; ages between 9 months and 4 years, 11 months and 29 days old; 18 years to 50 years old
  Interventions: Biological: yellow fever vaccine

INTERVENTIONS:
Biological: yellow fever vaccine — yellow fever vaccination in naive individuals who leaves in a state where this type of vaccination is not recommendated

SUMMARY:
The study main objective is to assess the immune status of children and adults who have never vaccinated, they will receive the first dose of 17DD yellow fever vaccine provided by the study and will be monitored for 10 years. Depending on the results of the analyzed of the data, the period of monitoring may be extended.

DETAILED DESCRIPTION:
This is a Phase IV study cohort, uncontrolled, composed of two segments: children and healthy adults. It will be included 2756 children and 2005 adults, evaluated initially in six different times (before vaccination, 30-45 days, 1 year, 4 years, 7 years and 10 years after vaccination). The Paraiba state was selected for the study because in this region there are no yellow fever virus dissemination and therefore no NIP recommendation for people's routine vaccination. However, the NIP indicate yellow fever vaccination for individuals who are moving to areas with virus circulation. The study will take place in six (6) Basic Health Units of three (3) municipalities (2 units per municipality) in the state of Paraíba. The selected municipalities are: Alhandra, Caaporã and Conde. The study target population consisted of healthy children and adults of both sexes. Children must be between 9 months and 4 years,11months and 29 days; adults between 18 and 50 years. It will be eligible for the study, people who have never received the yellow fever vaccine checked in vaccine design and history and who agree to participate. Not be included participants with any contraindication to vaccination against yellow fever and individuals who previously moved to risk areas for extended periods.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and sign the Informed Consent Term
2. Acceptance in participate on the study after reading, understanding and signed the Informed Consent Term
3. Participants of both sexes aged 9-4 years, 11 months and 29 days, after it was provided they have not received or have to receive the MMR or Tetraviral vaccine within 30 days or less.
4. Healthy adults of both sexes aged between 18 and 50 years since they have not received or have to receive the MMR or Tetraviral vaccine within 30 days or less.
5. Residence fixed in the municipality where the Basic Health Unit will held vaccination and collection of biological material samples (blood) for the study at the time of participant enrollment.
6. Availability to follow the proposed activities throughout the study period.
7. Agreement to provide name, address, telephone number and other information for personal contact is possible, if necessary (for example, event of failure to visit scheduled for follow-up).
8. Availability to follow the study protocol.
9. Acceptance for serological testing for HIV.
10. In adult women, it will be conduct pregnancy test (TIG).
11. Being in good health with no significant medical history (such as those described in Exclusion criteria).
12. Physical examination of screening with no significant clinical changes.

Exclusion Criteria:

1. Previous vaccination against yellow fever.
2. Presumed or confirmed pregnancy at any stage.
3. Women who are breastfeeding.
4. People in use, or have made use of immunosuppressants medicines.
5. People with personal history of anaphylactic reaction to food, drugs or vaccines.
6. People with personal history of allergy to egg ,erythromycin, kanamycin or gelatin.
7. People with autoimmune diseases.
8. Individuals seropositive for HIV.
9. People with thymic disease history, such as thymoma, myasthenia due to thymectomy and thymoma.
10. People who have received immunoglobulin, blood transfusions or derivatives in the last 60 days.
11. People who have received live virus vaccines or against cholera in the last 30 days, or who plan to receive them within 30 days after vaccination against yellow fever.
12. Individuals who have resided in an endemic area.
13. People with acute febrile disease and a compromised general health.
14. People immunosuppressed by disease (eg, cancer, AIDS, HIV infection with impaired immunity, etc.) or drugs (immunosuppressive drugs, radiotherapy, etc.).

Ages: 9 Months to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4761 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Immune response evolution in children and adults for yellow fever vaccine | before vaccination (day 0)
  seropositivity proportion and the yellow fever neutralizing antibodies geometric mean titers.
Immune response evolution in children and adults for yellow fever vaccine | 30-45 days after vaccination
  seropositivity proportion and the yellow fever neutralizing antibodies geometric mean titers.
Immune response evolution in children and adults for yellow fever vaccine | 1 year after vaccination
  seropositivity proportion and the yellow fever neutralizing antibodies geometric mean titers.
Immune response evolution in children and adults for yellow fever vaccine | 4 years after vaccination
  seropositivity proportion and the yellow fever neutralizing antibodies geometric mean titers.
Immune response evolution in children and adults for yellow fever vaccine | 7 years after vaccination
  seropositivity proportion and the yellow fever neutralizing antibodies geometric mean titers.
Immune response evolution in children and adults for yellow fever vaccine | 10 years after vaccination
  seropositivity proportion and the yellow fever neutralizing antibodies geometric mean titers.

SECONDARY OUTCOMES:
Interaction between dengue antibodies and the immune response evolution for yellow fever vaccine in children and adults. | before vaccination (day 0)
  Anti-dengue virus IgG antibodies and neutralizing antibodies to yellow fever vaccine.
Interaction between dengue antibodies and the immune response evolution for yellow fever vaccine in children and adults. | 30-45 days after vaccination
  Anti-dengue virus IgG antibodies and neutralizing antibodies to yellow fever vaccine.
Interaction between dengue antibodies and the immune response evolution for yellow fever vaccine in children and adults. | 1 year after vaccination
  Anti-dengue virus IgG antibodies and neutralizing antibodies to yellow fever vaccine.
Association between sociodemographic factors, personal medical history and immune status to yellow fever in children and adults | immediately before vaccination ( day 0 )
  Number of vaccine doses, age of the participant per years, age at vaccination, gender, personal vaccination record, vaccination history against yellow fever in infants' mothers, history of severe diseases (hospitalization, sequels, disability ), comorbidities and medications used at the time of blood collection.
Association between sociodemographic factors, personal medical history and immune status to yellow fever in children and adults | 1 year after vaccination
  Number of vaccine doses, age of the participant per years, age at vaccination, gender, personal vaccination record, vaccination history against yellow fever in infants' mothers, history of severe diseases (hospitalization, sequels, disability ), comorbidities and medications used at the time of blood collection.
Association between sociodemographic factors, personal medical history and immune status to yellow fever in children and adults | 4 years after vaccination
  Number of vaccine doses, age of the participant per years, age at vaccination, gender, personal vaccination record, vaccination history against yellow fever in infants' mothers, history of severe diseases (hospitalization, sequels, disability ), comorbidities and medications used at the time of blood collection.
Association between sociodemographic factors, personal medical history and immune status to yellow fever in children and adults | 7 years after vaccination
  Number of vaccine doses, age of the participant per years, age at vaccination, gender, personal vaccination record, vaccination history against yellow fever in infants' mothers, history of severe diseases (hospitalization, sequels, disability ), comorbidities and medications used at the time of blood collection.
Association between sociodemographic factors, personal medical history and immune status to yellow fever in children and adults | 10 years after vaccination
  Number of vaccine doses, age of the participant per years, age at vaccination, gender, personal vaccination record, vaccination history against yellow fever in infants' mothers, history of severe diseases (hospitalization, sequels, disability ), comorbidities and medications used at the time of blood collection.
Immune response evolution in children and adults for yellow fever vaccine that did not respond to the first dose and were revaccinated. | Immediately before vaccination
  seropositivity proportion and the yellow fever neutralizing antibodies geometric mean titers.
Immune response evolution in children and adults for yellow fever vaccine that did not respond to the first dose and were revaccinated. | 30-45 days after revaccination
  seropositivity proportion and the yellow fever neutralizing antibodies geometric mean titers.
Immune response evolution in children and adults for yellow fever vaccine that did not respond to the first dose and were revaccinated. | 1 year after first vaccination
  seropositivity proportion and the yellow fever neutralizing antibodies geometric mean titers.
Immune response evolution in children and adults for yellow fever vaccine that did not respond to the first dose and were revaccinated. | 4 years
  seropositivity proportion and the yellow fever neutralizing antibodies geometric mean titers.
Immune response evolution in children and adults for yellow fever vaccine that did not respond to the first dose and were revaccinated. | 7 years after first vaccination
  seropositivity proportion and the yellow fever neutralizing antibodies geometric mean titers.
Immune response evolution in children and adults for yellow fever vaccine that did not respond to the first dose and were revaccinated. | 10 years after first vaccination
  seropositivity proportion and the yellow fever neutralizing antibodies geometric mean titers.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Sergio S Sousa, MD, Principal Investigator — Universidade Federal da Paraíba
Locations (6):
- Brazil (6):
  - Unidade de Saúde da Família Oiteiro I, Alhandra, Paraíba
  - Unidade Saúde da Família Mata Redonda 1, Alhandra, Paraíba
  - Unidade de Saúde da Família Cupissura I, Caaporã, Paraíba
  - Unidade de Saúde da Família Santo Antônio, Caaporã, Paraíba
  - Unidade de Saúde da Família N Sra da Conceição, Conde, Paraíba
  - Unidade de Saúde da Família N Sra das Neves, Conde, Paraíba